CLINICAL TRIAL: NCT04013581
Title: Quadruple Oral Combination Therapy for Type 2 Diabetes Mellitus : Glycemic Control by Thiazolidinedione (TZD) or Sodium Glucose Co-transporter 2 (SGLT-2) Inhibitor as an add-on Therapy in Type 2 Diabetes Mellitus After Failure of an Oral Triple Antidiabetic Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0393
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Prospective, open label, randomized, parallel, multicenter clinical trial
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TZD group (Experimental): Pioglitazone added to Metformin, DPP-4 inhibitors, Sulfonylurea
  Interventions: Drug: TZD group
- SGLT-2 inhibitor group (Active Comparator): Empagliflozin added to Metformin, DPP-4 inhibitors, Sulfonylurea
  Interventions: Drug: SGLT-2 group

INTERVENTIONS:
Drug: TZD group — Pioglitazone 15mg (Acpio®, once daily, regardless of meal time, for 24 weeks) will be added for T2DM(type 2 diabetes mellitus) patients who had inadequate glycemic control (7% <HbA1c ≤ 10%) with triple therapy (metformin, DPP-4 inhibitors, sulfonylurea). At visit 3 (after 12 week-treatment), patients whose HbA1c level is more than 7.0% will be prescribed increased dosage of pioglitazone : from 15mg to 30mg
  Other Names: Acpio
  Arms: TZD group
Drug: SGLT-2 group — Empagliflozin 10mg (Jardiance®, once daily, regardless of meal time, for 24 weeks) will be added for T2DM patients who had inadequate glycemic control (7% <HbA1c ≤ 10%) with triple therapy (metformin, DPP-4 inhibitors, sulfonylurea). At visit 3 (after 12 week-treatment), patients whose HbA1c level is more than 7.0% will be prescribed increased dosage of empagliflozin : from 10mg to 25mg
  Other Names: Jardiance
  Arms: SGLT-2 inhibitor group

SUMMARY:
In the treatment of type 2 diabetes (T2D), the number of patients requiring combination therapy of oral antidiabetic agents (OADs) is more than 70%. Especially in Korea, the tendency to avoid insulin therapy is relatively higher than other countries, therefore, the need for combination therapy of OADs is quite high. However, according to the current guidelines, clinicians are recommended to prescribe three or fewer OADs as the combination therapy for T2D. Recently, various OADs have been developed, and it is expected that quadruple combination therapy of OADs would be quite effective to lower blood glucose levels. In the present study, the investigators designed the study to compare the efficacy and safety of quadruple combination therapy; thiazolidinedione (TZD) vs. SGLT-2 inhibitor as an add-on therapy to triple combination therapy (Metformin, Sulfonylurea, Dipeptidyl peptidase-4(DPP-4) inhibitors). Quadruple combination therapy group with the SGLT-2 inhibitor will be considered as active control group, because it have shown non-inferior glycemic efficacy to the conventional insulin conversion therapy in a previous clinical study. Patients who could not achieve the target blood glucose level (7% <HbA1c ≤ 10%) under the triple combination therapy (Metformin, Sulfonylurea, DPP-4 inhibitors) for more than 12 weeks will be enrolled in this prospective, open-label, randomized, parallel comparison, multicenter clinical trial. Subjects in each group (60 patients/group) will be treated with TZD-containing quadruple therapy or SGLT-2 inhibitor-containing quadruple therapy for 24 weeks. The investigators will evaluate the glycemic efficacy and safety of each group. Primary outcome is the 24 week-change of HbA1c from baseline levels.

ELIGIBILITY:
Inclusion Criteria:

* 1. 19 ≤ age ≤ 80, male or female
* 2. Type 2 diabetes patients who have taken triple combination therapy of OADs as followed : Metformin (≥1000 mg/day), Sulfonylurea (Glimepiride ≥ 4 mg/day or Gliclazide ≥ 60 mg/day), DPP-4 inhibitor (Full dose) for over 12 weeks
* 3. At screening, 7% < HbA1c ≤ 10%
* 4. Patients who refused insulin therapy.
* 5. Subjects who understood the contents of the clinical trial and are cooperative in the trial progress, and are considered to be able to participate until the end of the trial.
* 6. Patients who have voluntarily agreed in writing to participate in the clinical trial after hearing the explanation of the trial.

Exclusion Criteria:

* 1. Type 1 diabetes, gestational diabetes, and other types of diabetes than type 2 diabetes mellitus.
* 2. Patients who have the history of allergy of hypersensitivity for the medication of the clinical trial.
* 3. Patients who have the history of taking TZDs or SGLT-2 inhibitors within a year prior to screening visit, or have the history of discontinuation of them due to severe side effects.
* 4. Patients who have the history of acute or chronic metabolic acidosis including diabetic ketoacidosis (with or without coma), or any kinds of ketosis within 12 weeks prior to screening visit.
* 5. Patients who have genetic metabolic diseases, such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* 6. Patients who have the history of taking steroids for more than 2 weeks, within 8 weeks prior to screening visit.
* 7. Patients who have the history of malignancy within 5 years prior to screening visit (In case of bladder cancer, subjects will be excluded regardless of the time of diagnosis)
* 8. Patients who have the history of coronary artery bypass surgery or percutaneous coronary intervention, or suffered from heart failure (NYHA class III, IV)
* 9. Patients who have the history of uncontrolled arrhythmia, unstable angina, myocardial infarction, stroke, transient ischemic attacks, and cerebral vascular disease within 24 weeks prior to the screening date.
* 10. Patients of chronic renal failure, chronic kidney disease stage 3~5 (estimated glomerular filtration rate calculated vial CKD-EPI <60 mL/min/1.73m2) or on dialysis therapy.
* 11. Elevated liver enzymes (AST, ALT, ALP ≥ 2.5*upper limit of normal (ULN) or Total bilirubin ≥ 2.5*ULN) or Child-Pugh class B or C (for the patients of liver cirrhosis)
* 12. Subjects who are pregnant or lactating
* 13. Perioperative patients, patients with severe infections or severe trauma
* 14. Patients with unexamined gross hematuria
* 15. Any other subjects who is determined to be ineligible for the clinical trials by researchers.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c | 12 weeks
Change of HbA1c | 24 weeks
  Mean difference of HbA1c after 24 week-treatment

SECONDARY OUTCOMES:
glucose | 12 weeks
  Percentage of patients who achieve target HbA1c (≤7% level)
glucose | 24 weeks
  Mean difference of fasting blood glucose after 24 week-treatment
Adverse events | 12 weeks
  Incidence of adverse events during treatment period
Adverse events | 24 weeks
  Incidence of adverse events during treatment period
Change of kidney function | 12 weeks
  Mean change of BUN and serum creatinine
Change of kidney function | 24 weeks
  Mean change of BUN and serum creatinine
Change of liver enzymes | 12 weeks
  Mean change of AST(Asparate aminotransferase)
Change of liver enzymes | 12 weeks
  Mean change of ALT(Alanine aminotransferase)
Change of liver enzymes | 12 weeks
  Mean change of Total bilirubin
Change of liver enzymes | 24 weeks
  Mean change of AST
Change of liver enzymes | 24 weeks
  Mean change of ALT
Change of liver enzymes | 24 weeks
  Mean change of Total bilirubin

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No